CLINICAL TRIAL: NCT00722020
Title: High Frequency Chest Wall Oscillation in Hospital Management of Asthmatic Children
Brief Title: HFCWO in Hospitalized Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-0078
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Bronchial Asthma; Asthma; Status Asthmaticus
Keywords: Asthma; Bronchial Disease; Status Asthmaticus; High Frequency Chest Wall Oscillation; the Vest; HFCWO
MeSH Terms: conditions — Asthma; Status Asthmaticus; Bronchial Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vest Arm (Experimental): HFCWO treatments 2-3 times daily 15 minutes per treatment via the VEST
  Interventions: Device: VEST
- Control (No Intervention): Historical control for PICU asthma patients

INTERVENTIONS:
Device: VEST — 15 minutes of HFCWO via the Vest 2-3 times daily
  Other Names: Hill-Rom Vest(tm)
  Arms: Vest Arm

SUMMARY:
To determine whether or not high frequency chest wall oscillation (in the form of the VestTM) is superior to regular asthma therapy in the management of children hospitalized with moderate to severe asthma.

DETAILED DESCRIPTION:
A historically controlled pilot study was conducted in pediatric patients 18 months to 18 years of age hospitalized with a diagnosis of asthma or reactive airway disease and admitted to the pediatric intensive care unit. Upon receiving informed consent, patients were treated with HFCWO therapy via the VEST. The primary endpoint was time to readiness for discharge, lack of need for continued supportive care (e.g., intravenous fluid or oxygen), and bronchodilator treatments spaced at least four hours apart.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric patient between the ages of 18 months and 18 years admitted to Winthrop University Hospital's pediatric floor or intensive care unit with a diagnosis of asthma or reactive airway disease

Exclusion Criteria:

* Patients with chronic, comorbid respiratory conditions (e.g., cerebral palsy, cystic fibrosis)
* Those who regularly use HFCWO
* Any patient exhibiting an absolute contraindication to HFCWO therapy
* Absolute contraindications to using HFCWO include head and neck injury prior to stabilization, and active hemorrhage with hemodynamic instability

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Roberts, MD, Principal Investigator — Winthrop University
Locations (2):
- United States (2):
  - Winthrop University Hospital, Winthrop Pediatric Associates, Long Island City, New York
  - Winthrop University Hospital, Long Island City, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- HFCWO / VEST Group: Patients will receive HFCWO therapy via the VEST(TM). Each Vest treatment will be accompanied by a simultaneous nebulized bronchodilator treatment.
  High Frequency Chest Wall Oscillation via Vest (Hill-Rom Vest(tm)): Simultaneous to bronchodilator treatment via nebulizer (regular treatment), patients will receive 15 minutes of HFCWO via the Vest.
- Standard Care: Regular nebulized bronchodilator treatment. Sham Vest treatment as investigator is blinded to whether patient actually received Vest treatment.
  Regular nebulized bronchodilator treatment.: Sham Vest treatment.
Period: Overall Study
Arm/Group | HFCWO / VEST Group | Standard Care
Started | 19 | 24
Completed | 19 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pediatric patients admitted with diagnosis of Asthma
Groups:
- HFCWO / VEST: Pediatric patients with primary diagnosis of Asthma received HFCWO therapy via the VEST(TM). Each Vest treatment will be accompanied by a simultaneous nebulized bronchodilator treatment. Patients receive 15 minutes of HFCWO via the Vest.
- Standard Care With Sham Vest: Regular nebulized bronchodilator treatment. Sham Vest treatment as investigator is blinded to whether patient actually received Vest treatment.
- Total: Total of all reporting groups
Arm/Group | HFCWO / VEST | Standard Care With Sham Vest | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (2.3) | 8.2 (2.0) | 8.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be Time to Readiness for Discharge.
Description: Days in the hospital prior to patient being clinically ready to discharge
Time Frame: 30 days
Population: asthmatic children
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HFCWO / VEST Group | Standard Care
Number analyzed (Participants) | 19 | 24
days | 1.74 (.7) | 1.75 (.6)

2. Secondary Outcome: Secondary Endpoint Total Hospital Length of Stay
Description: Seconadary endpoint was Total Hospital length of stay
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HFCWO / VEST | Standard Care With Sham Vest
Number analyzed (Participants) | 19 | 24
days | 2.5 (0.8) | 2.5 (0.7)

ADVERSE EVENTS:
Time Frame: ICU admission and hospital admission time
Arm/Group | HFCWO / VEST | Standard Care With Sham Vest
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/24
Other Adverse Events (participants affected / at risk) | 0/19 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No